CLINICAL TRIAL: NCT00480766
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, 12-Month Study to Evaluate the Efficacy and Safety of Oral Alendronate Sodium Once Weekly for the Prevention and Treatment of Glucocorticoid-Induced Bone Loss
Brief Title: A Research Study to Evaluate the Safety and Effectiveness of MK0217 to Prevent and Treat Bone Loss (0217-193)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0217-193; 2007_560
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis
Keywords: Glucocorticoid
MeSH Terms: conditions — Osteoporosis | interventions — Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0217/Duration of Treatment : 12 Months

SUMMARY:
A research study to see how safe and effective MK0217 is when taken weekly for the prevention and treatment of steroid induced bone loss.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 to 80 years, being treated with oral glucocorticoid (steroid), without vertebral fracture or prior osteoporotic fracture

Exclusion Criteria:

* Mentally or legally incompetent, pregnant, alcohol or drug dependence, history of heart disease, kidney disease, hypertension, upper gastrointestinal disease, cancer, being treated with hormone replacement therapy, or life expectancy of less than 3 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2001-07; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Assess the effect of patients taking MK0217 once weekly along with steroids for a 12 month period by checking the percentage change of bone mineral density as compared to patients taking placebo

SECONDARY OUTCOMES:
Describe how safe and tolerable the drug MK0217 is when patients take it once weekly over 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Stoch SA, Saag KG, Greenwald M, Sebba AI, Cohen S, Verbruggen N, Giezek H, West J, Schnitzer TJ. Once-weekly oral alendronate 70 mg in patients with glucocorticoid-induced bone loss: a 12-month randomized, placebo-controlled clinical trial. J Rheumatol. 2009 Aug;36(8):1705-14. doi: 10.3899/jrheum.081207. Epub 2009 Jun 1. PMID 19487264